CLINICAL TRIAL: NCT04064138
Title: Erector Spinea Plane Block Versus Peritoneal Block Analgesia in Laparoscopic Cholecystectomy
Brief Title: Analgesic Effect of Erector Spinea Plane Block Compared to Peritoneal Block in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MS ∕ 19.01.436
Record Dates: First submitted 2019-07-12; First posted 2019-08-21 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2019-12

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant
Masking Description: - Single blind (participant) study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peritoneal block (Active Comparator): patients will receive peritoneal block as an adjuvant analgesic technique.
  Interventions: Procedure: Peritoneal block; Other: General anesthesia
- Ultrasound guided erector spinae plane block (Active Comparator): Patients will receive ultrasound guided erector spinae plane block
  Interventions: Procedure: Ultrasound guided erector spinae plane block; Other: General anesthesia

INTERVENTIONS:
Procedure: Peritoneal block — At the beginning of surgery, immediately after insertion of the first port 2 mg/kg lidocaine and 25mg/kg magnesium sulfate and 1/200 000 epinephrine in a total volume 50 ml (completed with saline .9%) will be given intra-peritoneal 10 min before the surgeon proceeds . At the end of the surgery another similar lidocaine-magnesium-epinephrine injection will be instillated before removal of the last port and the drain will be kept closed for 30 min.
  Arms: Peritoneal block
Procedure: Ultrasound guided erector spinae plane block — Before general anesthesia, ESPB will be performed under ultrasound guidance. The linear ultrasound transducer will be placed in a longitudinal parasagittal orientation 3 cm lateral to the T9 spinous process. The erector spinae muscles will be identified superficial to the tip of the T9 transverse process. The patient's skin will be anesthetized with 3 mL of 2% lidocaine. A 21 gauge 10cm needle will be inserted using an in plane superior to inferior. The tip of the needle will be placed into the facial plane on the deep aspect of erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting erector spinae muscle off the bony shadow of the transverse process on ultrasonographical imaging. The calculated dose of lidocaine (2mg/kg) with 150 mg MgSo4 and 1/200 000 epinephrine will be injected on each side.
  Arms: Ultrasound guided erector spinae plane block
Other: General anesthesia — General anesthesia

SUMMARY:
The aim of this study is to detect weather peritoneal block or erector spinae plane block will provide the most ideal analgesia for patients undergoing laparoscopic cholecystectomy. Peritoneal block by instillation of local anesthetic into the peritoneal cavity will act by blocking the free afferent nerve endings in the peritoneum and the systemic absorption of local anesthetic from the peritoneal cavity may also play a part in reduced pain.

On the other hand ,the erector spinae plane block is a novel analgesic technique that provide both visceral and somatic analgesia due to its communication with the paravertebral space. Local anesthetic mixture of lidocaine , magnesium sulphate and epinephrine will be used for both techniques.

DETAILED DESCRIPTION:
The pain that a patient feels after laparoscopic cholecystectomy results from three different and clinically separate components: somatic pain due to trocar insertion sites , visceral pain due to surgical dissection and tissue handling at the gall bladder bed, and shoulder pain due to retention of carbon dioxide in the abdomen, which irritates the phrenic nerve and diaphragm. Ineffective treatment of post laparoscopic cholecystectomy pain may delay recovery and mandate inpatient admission and therapy and increase the cost of such care.

The aim of this study is to evaluate the analgesic effect of Erector spinea plane block in comparison with peritoneal block for laparoscopic cholecystectomy. Serum level of cortisol as a stress biomarker ,perioperative primary hemodynamics ,visual analogue scale , patient request for rescue analgesia and occurrence of side effects are the parameters for comparison between both techniques. Each patient will be followed up for 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* American physical status classes I and II

Exclusion Criteria:

* Patient refusal.
* Pregnancy
* Neuromuscular diseases (as myopathies, myasthenia gravies…)
* Hematological diseases.
* Bleeding diseases.
* Coagulation abnormality.
* Psychiatric diseases.
* Local skin infection at site of the block.
* Local skin sepsis at site of the block.
* Known intolerance to the study drugs.
* Body Mass Index > 40 Kg/m2.
* Chronic renal disease.
* Chronic hepatic disease.
* Preexisting neurological deficit.
* Conversion to open cholecystectomy
* Excessively long surgical times (> 90 min)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Time for first requirement of rescue analgesia | for 24 hours after surgery
  an analgesic (nalbuphine 10 mg ) will be administer postoperatively on patient request in case of the pain score ≥ 4/10 on VAS. It represent the end point of the study which determines the duration of analgesia

SECONDARY OUTCOMES:
Peripheral oxygen saturation | one hour before induction general anesthesia then every 10 min till end of surgery then every 4 hours till end of first 24 hours.
  estimate of oxygenated hemoglobin concentration in the blood , measured by pulse oximeter device
mean arterial blood pressure | one hour before induction general anesthesia then every 10 min till end of surgery then every 4 hours till end of first 24 hours.
  The average pressure in the arteries during one cardiac cycle.
heart rate | one hour before induction general anesthesia then every 10 min till end of surgery then every 4 hours till end of first 24 hours.
  Number of heart beats per minute. Lower heart rate implies better cardiovascular fitness and less stress.
end tidal CO2 | immediately after intubation and ever 10 min till the end of surgery.
  amount of carbon dioxide in each breathe .
Intensity of Abdominal Pain: visual analogue scale | immediately after recovery ,then every 4 hours for 24 hour.
  Postoperative assessment of abdominal pain using visual analogue scale (1-10), where 1 equals no pain and 10 indicates the worst possible pain.
Intensity of Shoulder Pain: five point scale | immediately after recovery ,then every 4 hours for 24 hour.
  shoulder pain score scale:
  1. no pain( the best outcome)
  2. discomfort in shoulder but no pain
  3. light pain ( analgesia not required)
  4. moderate pain ( analgesia required)
  5. sever pain ( analgesia and sedation required ) (the worst outcome)
serum cortisol level | preoperative and one hour postoperative.
  a steroid hormone secreted from adrenal cortex in response to stress.
Post-operative total analgesic requirement | for 24 hours postoperatively.
  total amount of nalbuphine consumed by the patient from the time of first analgesic requirement till the end of 24 hours.
nausea | immediately after recovery and every 4 hours for 24 hour postoperatively
  four point verbal rating score to assess the incidence of nausea and vomiting where 1 indicate they did not happen , 2 indicate nausea and 3 indicate vomiting for once and 4 indicate repeated vomiting
vomiting | immediately after recovery and every 4 hours for 24 hour postoperatively
  four point verbal rating score to assess the incidence of nausea and vomiting where 1 indicate they did not happen , 2 indicate nausea and 3 indicate vomiting for once and 4 indicate repeated vomiting.
dizziness | immediately after recovery and every 4 hours for 24 hour postoperatively
  a questionnaire will be collected to detect the incidence of occurrence of dizziness
tinitus | immediately after recovery and every 4 hours for 24 hour postoperatively
  a questionnaire will be collected to detect the incidence of occurrence of tinnitus
circumoral numbness | immediately after recovery and every 4 hours for 24 hour postoperatively
  a questionnaire will be collected to detect the incidence of occurrence of circumoral numbness

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Sultan, MD, Study Chair — Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Central Hospital, gastroenterology surgery centre, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
1. individual participant data will be available.
  2. all individual participant data collected during the trial after deidentification will be shared.
  3. The data will be shared with anyone who wishes to access the data for any purpose .
Supporting Information: Study Protocol, SAP, ICF
Time Frame: data will be available immediately following publication with no end date
Access Criteria: 1. individual participant data will be available.
  2. all individual participant data collected during the trial after deidentification will be shared.
  3. study protocol, statistical analysis and informed consent form will be available.
  4. data will be available immediately following publication with no end date.
  5. the data will be shared with anyone who wishes to access the data for any purpose.
  6. data will be available at www.researchgate.net/profile/Sameh_Ghareeb3
URL: http://www.researchgate.net/profile/Sameh_Ghareeb3